CLINICAL TRIAL: NCT06546033
Title: Determination of the Effects of Intermittent Fasting and Mediterranean Diet on Quality of Life, Circadian Rhythm and Appetite Markers in Patient With Multiple Sclerosis
Brief Title: Intermittent Fasting and Mediterranean Diet in Patient With Multiple Sclerosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nigde Omer Halisdemir University (Other)
Collaborators: Acibadem University (Other)
Responsible Party: Principal Investigator, Elif Gökçe İNBAŞI, Lecturer, MSc., Nigde Omer Halisdemir University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-7/286
Record Dates: First submitted 2024-07-30; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Multiple Sclerosis; Intermittent Fasting
Keywords: Multiple sclerosis; circadian rhythm; mediterranean diet; Intermittent Fasting
MeSH Terms: conditions — Multiple Sclerosis; Intermittent Fasting

STUDY DESIGN:
Intervention Model Description: The first group will be fed with Mediterranean diet The second group will be fed with intermittent diet
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1. Group (intermittent fasting) (Experimental): Time Restricted Diet (10.00-18.00)
  Interventions: Other: application of different types of diet
- 2. Group (mediterranean diet) (Experimental): Diet based on the consumption of plant foods, cereals, oilseeds, etc.
  Interventions: Other: application of different types of diet

INTERVENTIONS:
Other: application of different types of diet — application of different types of diet

SUMMARY:
When the literature was reviewed, there is no study in which the effects of intermittent fasting and Mediterranean diet on quality of life, sleep, circadian rhythm and appetite hormones leptin and ghrelin levels in MS patients were evaluated and the two diet types were comparatively examined in terms of all these parameters.

DETAILED DESCRIPTION:
Multiple Sclerosis (MS) is the most common chronic inflammatory disease affecting young adults between the ages of 20-40 years, which causes irreversible neurological damage and symptoms and is influenced by genetic and environmental factors on the Central Nervous System. Depression that may occur in MS patients leads to decreased motivation and negatively affects the quality of life. At the same time, depression may be accompanied by sleep disorders, anxiety, fatigue and eating disorders. Nutrition is recognised as one of the possible risk factors for the development of MS and has potential applications in the management and treatment of the disease. When the literature was reviewed, there is no study evaluating the effect of intermittent fasting and Mediterranean diet on quality of life, sleep, circadian rhythm and appetite hormones leptin and ghrelin levels in MS patients and comparing the two diet types in terms of all these parameters.

ELIGIBILITY:
Inclusion Criteria:

* To apply to the neurology outpatient clinic, to be a female between the ages of 18-65 who has been diagnosed with MS by a physician
* Not being in the attack period
* Not being in menopause Not being diagnosed with any autoimmune system disease other than -MS that may adversely affect the study,
* Not following the Mediterranean diet and intermittent fasting programmes in the last three months,
* Not being diagnosed with an eating behaviour disorder,
* Not having any communication problems,
* Signing the informed consent form,
* Brain MRI within the last three months,
* Not to be pregnant and lactating
* No physical disability No history of cancer
* Body Mass Index between 18,5 kg/m2- 29,9 kg/m2,
* Not losing 5% and/or more body weight in the last month

Exclusion Criteria:

* Having a diagnosis of autoimmune system disease that may adversely affect working outside of -MS,
* To be in the attack period-Being under 18 years of age and over 65 years of age
* Being in menopause-Mediterranean diet and intermittent fasting feeding programmes within the last three months,
* Diet therapy that has an effect on the autoimmune system within the last three months,
* Being diagnosed with eating behaviour disorder,
* Having any communication problems,- Not signing the informed consent form,
* Failure to adapt to the work during the working period, to be in a situation/behaviour that may adversely affect the work,
* To have applied any nutritional intervention during the last three months prior to the study,
* Taking supplements such as selenium, zinc, iron, vitamin D and/or B12, which may affect the course of the study,
* To have received cancer treatment and / or to be receiving cancer treatment,
* Other neurological diseases (e.g. Parkinson's, epilepsy, Alzheimer's),
* Diagnosed with a disease lasting more than 4 months in the last 12 months and other specialised dietary / compositionally different dietary patterns (e.g. high protein, ketogenic, low energy content < 1000 kcal/day),
* Body Mass Index <18.5 kg/m2 or >30 kg/m2
* Losing 5% and/or more body weight in the last month,
* Having a physical disability

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-05-02 (Actual); Primary Completion 2026-09-02 (Estimated); Study Completion 2026-12-02 (Estimated)

PRIMARY OUTCOMES:
Biochemical parameter | baseline- 3 months
  Hemogram values of the group 1 and group 2 patients with multiple sclerosis participating in the study will be compare.

SECONDARY OUTCOMES:
The Morning and Evening Questionnaire | baseline- 3 months
  The Morning and Evening Questionnaire was developed by Horne and Ostberg in 1975. The Turkish validity and reliability scale has 19 questions and is unidimensional. It is a 5-point Likert type (1=absolutely morning person-5=absolutely evening person) and the score that can be obtained from the scale varies between 0 and 86. Each score to be taken from the scale remains in different score ranges. This represents a different personality trait.
Pittsburgh Sleep Quality Index | baseline- 3 months
  Pittsburgh Sleep Quality Index (PSQI) was developed by Buysse et al. The scale, which was developed by Buysse et al. and its Turkish validity and reliability was performed, consists of 18 self-report questions and measures the sleep quality of the individual in the last 4 weeks. PDQI has 7 components. Each of these components is scored between 0-3. A minimum score of 0 and a maximum score of 21 is obtained from the scale. A total score of 5 and above indicates poor sleep quality.
Multiple Sclerosis Quality of Life-MuSiQoL | baseline- 3 months
  Multiple Sclerosis Quality of Life-MuSiQoL scale was developed by Vickrey et al. in 1995 to evaluate the quality of life of MS patients. The original version consists of 74 questions and there is also a short form consisting of 31 questions. MuSiQoL consists of a total of 9 subgroups including activities of daily living, psychological status, findings, friendships, family relationships, emotional and sexual life, acceptance, coping with the disease and satisfaction with health services. During the assessments, individuals are asked to answer by taking into account their situation in the last 4 weeks. They are asked to tick the option that best expresses themselves from the options of never (0: Never), rarely (1: Occasionally), sometimes (2: Some), frequently (3: Very) and always (4: Very much). Turkish validity and reliability studies were conducted.

CONTACTS AND LOCATIONS:
Overall Officials: Nihan Çakır Biçer, PhD., Study Director — Acıbadem Mehmet Ali Aydınlar University
Locations (1):
- Nigde Omer Halisdemir University, Niğde, Bor, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No